CLINICAL TRIAL: NCT01041417
Title: Granulocyte-Macrophage Stimulating Factor (GM-CSF) and Mobilization of Progenitor Cells in Peripheral Arterial Disease: A Phase II Randomized Study
Brief Title: Granulocyte-Macrophage Stimulating Factor in the Treatment of Peripheral Arterial Disease
Acronym: GPAD-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00030362; 1RC2HL101515-01 (NIH)
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Arterial Disease
Keywords: claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GM-CSF (Experimental): Subjects will receive GM-CSF 500μg (Sargramostim (Leukine), Sanofi Aventis) by a self-administered subcutaneous injection thrice weekly on Monday, Wednesday, and Friday for four weeks
  Interventions: Drug: Granulocyte-Macrophage Stimulating Factor (GM-CSF)
- Placebo (Placebo Comparator): Subjects will receive a saline injection (placebo) by a self-administered subcutaneous injection thrice weekly on Monday, Wednesday, and Friday for four weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Granulocyte-Macrophage Stimulating Factor (GM-CSF) — 500 micrograms of GM-CSF
  Other Names: GM-CSF, Leukine
  Arms: GM-CSF
Drug: Placebo — Saline injection
  Arms: Placebo

SUMMARY:
Peripheral arterial disease is a common condition in older adults involving poor arterial circulation in the legs leading to leg pain and debility. The body's own circulating blood vessel stem cells may help to improve circulation. This study will test whether treatment with the drug granulocyte macrophage colony stimulating factor (GM-CSF) will improve symptoms and signs of peripheral arterial disease over placebo after four weeks of therapy. As well this study will examine whether improvements in blood vessel function can be observed. Finally, we will measure blood vessel function and stem cell levels in order to determine whether they can help to predict whether patients wither peripheral arterial disease will suffer further cardiovascular complications.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) affects more than 8 million Americans. Although exercise, smoking cessation, anti-platelet therapy, cilostazol, statins and revascularization are used to treat PAD, men and women with PAD have significantly greater functional impairment and fasterfunctional decline than those without PAD. Stem and progenitor cell (PC) therapy that promotes neoangiogenesis is an emerging treatment modality in PAD. Progenitor cells, particularly those of endothelial origin, are involved in vascular repair and regeneration. They originate primarily but not exclusively from the bone marrow, differentiate into endothelial and other vascular cells, and contribute to neovascularization during tissue repair by direct and paracrine mechanisms. Endogenous, pharmacologically-stimulated, and exogenous PCs contribute to re-endothelialization and neovascularization. Granulocyte colony stimulating factor (G-CSF) and granulocyte-macrophage colony stimulating factor (GM-CSF) stimulate mobilization of hematopoietic and other PCs from the bone marrow.In the murine hind limb ischemia model, GM-CSF administered by injection or by plasmid transfer augments circulating levels of PCs, increases capillary density, and promotes arteriogenesis.GM-CSF also augments neo-endothelialization of denuded arteries, promotes proliferation, differentiation and survival of hematopoietic cells, monocytes and macrophages.

ELIGIBILITY:
Inclusion Criteria:

* 160 males or post-menopausal females between 21 and 80 years of age. Female subjects must be (a) post-menopausal, (b) surgically sterile or (c) use adequate birth control and have a negative pregnancy test within 3 days prior to administration of study drug and should not be breastfeeding.
* Documented PAD (By Ankle-Brachial Indices or Angiographically)
* Clinically stable (at least 2 months) history of intermittent claudication with no change in symptom severity in the 2 months prior to screening.
* On stable statin therapy for previous 3 months.
* Peak Walking Time (PWT) between 1 and 12 minutes on a standardized Gardner treadmill protocol.
* A Doppler-derived ankle-brachial index (ABI) of < 0.85 in the symptomatic limb after 10 minutes of rest at screening. For subjects with an ABI of >1.3 (non-compressible arteries) a Toe-Brachial Index (TBI) of < 0.70 must be obtained for subject qualification, or if ABI is > 0.85 to 1.0 , and a reduction of 20% in ABI measured within 1 minute of treadmill testing.
* On appropriate and stable medical therapy for atherosclerosis for at least 2 months.
* Able to give informed consent.
* Diabetics with a dilated eye exam excluding proliferative retinopathy in the previous 12 months.

Exclusion Criteria:

* Recent or current active infections (treated with antibiotics).
* Recent (3 months) change in statin therapy
* Critical limb ischemia either chronic (category 3 and 4 of SVS classification) or acute ischemia manifested by rest pain, ulceration, or gangrene.
* Lower extremity vascular surgery, angioplasty or lumbar sympathectomy within 3 months of enrollment.
* Participation in a structured exercise treatment protocol within 3 months of enrollment.
* Prior myeloid cancer.
* Unstable angina, myocardial infarction, TIA, stroke or revascularization in the preceding 4 months.
* Severe heart failure (Class III or IV), heart muscle disease or atrial fibrillation.
* Limitation on exercise for symptoms other than intermittent claudication such as arthritis or dyspnea.
* Uncontrolled diabetes mellitus (defined as HbA1c > 10.0).
* Chronic renal disease (creatinine of >2.5 mg/dl) or hepatic disease (> 3 X elevations in AST and ALT).
* Ophthalmologic conditions associated with a neo-vascular response.
* Alcohol or drug abuse, or any other disease process that, in the opinion of the PI, will interfere with the ability of the patient to participate in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2009-09; Primary Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Poole J, Mavromatis K, Binongo JN, Khan A, Li Q, Khayata M, Rocco E, Topel M, Zhang X, Brown C, Corriere MA, Murrow J, Sher S, Clement S, Ashraf K, Rashed A, Kabbany T, Neuman R, Morris A, Ali A, Hayek S, Oshinski J, Yoon YS, Waller EK, Quyyumi AA. Effect of progenitor cell mobilization with granulocyte-macrophage colony-stimulating factor in patients with peripheral artery disease: a randomized clinical trial. JAMA. 2013 Dec 25;310(24):2631-9. doi: 10.1001/jama.2013.282540. PMID 24247554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2010 and July 2012, 322 individuals with peripheral artery disease were assessed for eligibility. 159 subjects were enrolled into the study from Emory Healthcare, Veterans Affairs hospitals in Atlanta, and Medical College of Georgia.
Groups:
- GM-CSF: Granulocyte-Macrophage Colony Stimulating Factor injection - three times for four weeks
  500 microgram dose of GM-CSF
- Placebo: Saline injection - three times for four weeks
Period: Overall Study
Arm/Group | GM-CSF | Placebo
Started | 80 | 79
Completed | 73 | 76
Not Completed | 7 | 3
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GM-CSF | Placebo | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (7.9) | 63.6 (7.9) | 63.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 70 | 69 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 34 | 79
  White | 33 | 45 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 80 | 79 | 159

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Walking Time During Treadmill Exercise Tolerance Test From Baseline to 3 Months
Description: Exercise Tolerance Test (ETT) was conducted using the Gardner protocol. Participants exercised on a treadmill, starting at 2.0 mph. The intensity of exercise (speed) was increased in grade of 2% every 2 minutes. Participants were asked to exercise until symptom limitation and the time measured in seconds from the ETT was used for data analysis.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
seconds | 109 (248) [67 to 151] | 56 (182) [14 to 98]

2. Secondary Outcome: Change in Peak Walking Time During Treadmill Exercise Tolerance Test From Baseline to 6 Months
Description: as for outcome 1
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
seconds | 112 [71 to 153] | 77 [36 to 117]

3. Secondary Outcome: Change in Claudication Onset Time (COT) From Baseline to 3 Months
Description: Claudication is pain, tired or weak feeling that occurs in the legs, usually during activity such as walking. The COT was measured as the time to onset of the participant's typical claudication as the maximum distance the patient could walk on the treadmill.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
seconds | 81 [52 to 111] | 61 [32 to 91]

4. Secondary Outcome: Change in Claudication Onset Time (COT) From Baseline to 6 Months
Description: as for outcome 3
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
seconds | 93 [64 to 122] | 61 [33 to 89]

5. Secondary Outcome: Change in Walking Distance Scores on Walking Impairment Questionnaire (WIQ) From Baseline to 3 Months
Description: The WIQ quantifies walking difficulty on a 100-point scale, in which 0 indicates extreme difficulty and 100 indicates no difficulty with walking distance.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- GM-CSF: Granulocyte-Macrophage Colony Stimulating Factor: 80 subjects were randomized to receive GM-CSF Monday, Wednesday and Friday for 4 weeks of therapy.
- Placebo: Placebo: 79 subjects were randomized to receive placebo on Monday, Wednesday and Friday for 4 weeks.
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 12.5 (27.6) [6.4 to 18.7] | 4.8 (24.8) [-0.2 to 9.8]

6. Secondary Outcome: Change in Walking Distance Scores on Walking Impairment Questionnaire (WIQ) From Baseline to 6 Months
Description: as for outcome 5
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 8.0 [2.1 to 14.0] | 3.7 [-0.9 to 8.3]

7. Secondary Outcome: Change in Walking Speed Score on Walking Impairment Questionnaire (WIQ) From Baseline to 3 Months
Description: The WIQ quantifies walking difficulty on a 100-point scale, in which 0 indicates extreme difficulty and 100 indicates no difficulty with walking speed.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 9.1 [4.2 to 14.0] | 7.5 [2.1 to 12.8]

8. Secondary Outcome: Change in Walking Speed Score on Walking Impairment Questionnaire (WIQ) From Baseline to 6 Months
Description: as for outcome 7
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 9.9 [4.6 to 15.3] | 8.5 [3.8 to 13.2]

9. Secondary Outcome: Change in Stair Climbing Score on Walking Impairment Questionnaire (WIQ) From Baseline to 3 Months
Description: The WIQ quantifies walking difficulty on a 100-point scale, in which 0 indicates extreme difficulty and 100 indicates no difficulty with stair climbing elements.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 8.5 [3.0 to 13.9] | 4.2 [-2.2 to 10.6]

10. Secondary Outcome: Change in Stair Climbing Score on Walking Impairment Questionnaire (WIQ) From Baseline to 6 Months
Description: as for outcome 9
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 10.4 [4.9 to 15.9] | 6.6 [1.2 to 11.9]

11. Secondary Outcome: Change in Score on Physical Composite Score (PCS) Subscale of the Short Form 36 Health Survey (SF-36) From Baseline to 3 Months
Description: The SF-36 is a standard quality of life instrument. The PCS represents the the physical burden on quality of life and is a summary of questions related to physical impact of a disease or condition (physical function, role physical, bodily pain, and general health). PCS is a summary measure derived from 8 scale score and the score ranges from 0-100; higher scores indicate better performance.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 4.1 [2.4 to 5.8] | 2.1 [0.5 to 3.7]

12. Secondary Outcome: Change in Score on Physical Composite Score (PCS) Subscale of the Short Form 36 Health Survey (SF-36) From Baseline to 6 Months
Description: as for outcome 11
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 5.2 [3.3 to 7.0] | 3.1 [1.5 to 4.7]

13. Secondary Outcome: Change in Score on Mental Composite Score (MCS) Subscale of the Short Form 36 Health Survey (SF-36) From Baseline to 3 Months
Description: The SF-36 is a standard quality of life instrument. The MCS represents the the mental burden on quality of life and is a summary of questions related to mental impact of a disease or condition (mental function, role emotional, vitality, and mental health). MCS is a summary measure derived from 8 scale score and the score ranges from 0-100; higher scores indicate better performance.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 0.7 [-1.5 to 2.9] | 2.4 [-0.2 to 5.0]

14. Secondary Outcome: Change in Score on Mental Composite Score (MCS) Subscale of the Short Form 36 Health Survey (SF-36) From Baseline to 6 Months
Description: as for outcome 13
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | -0.2 [-2.4 to 2.0] | 1.1 [-1.0 to 3.2]

15. Secondary Outcome: Change in Score on Physical Functioning Subscale of the Short Form 36 Health Survey (SF-36) From Baseline to 3 Months
Description: The SF-36 is a standard quality of life instrument. The physical functioning represents limitations in physical activities because of health problems. Physical functioning is a summary measure derived from 8 scale scores and the score ranges from 0-100; higher scores indicate better performance.
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 11.4 [6.7 to 16.1] | 4.8 [-0.1 to 9.6]

16. Secondary Outcome: Change in Score on Physical Functioning Subscale of the Short Form 36 Health Survey (SF-36) From Baseline to 6 Months
Description: as for outcome 15
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | GM-CSF | Placebo
Number analyzed (Participants) | 73 | 76
units on a scale | 14.3 [9.7 to 18.9] | 8.1 [3.7 to 12.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at weeks 1, 2, 3, 4, 8 and 3 month follow-up and 6 month follow-up
Groups:
- GM-CSF: Granulocyte-Macrophage Colony Stimulating Factor injection - Monday, Wednesday and Friday for 4 weeks of therapy.
  500 microgram dose of GM-CSF
- Placebo: Saline injection - Monday, Wednesday and Friday for 4 weeks.
Arm/Group | GM-CSF | Placebo
Serious Adverse Events (participants affected / at risk) | 9/80 | 9/79
Other Adverse Events (participants affected / at risk) | 79/80 | 69/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | GM-CSF (N=80) | Placebo (N=79)
Death (Social circumstances) | 1/73 (1) | 0/76 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Esophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain, non-cardiac (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Critical Limb Ischemia (Vascular disorders) | 1 (1) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elective Procedure (Surgical and medical procedures) | 1 (1) | 1 (1) — Admission for elective procedure
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Trauma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Admission for trauma
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF (N=80) | Placebo (N=79)
Headaches (Nervous system disorders) | 18 (18) | 9 (9)
Difficulty breathing (Cardiac disorders) | 5 (5) | 8 (8)
Chest pain (Cardiac disorders) | 6 (6) | 7 (7)
Joint/back/muscle pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 14 (14)
Gastrointestinal side effects (Gastrointestinal disorders) | 21 (21) | 11 (11)
Night sweats (General disorders) | 13 (13) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 41 (41) | 1 (1)
Swelling (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4)
Fatigue (General disorders) | 17 (17) | 9 (9)

LIMITATIONS AND CAVEATS:
Study population were subjects with claudication who underwent angiography. Study design could not show therapeutic benefit of GM-CSF therapy with dose and duration changes. And study design encouraged all subjects to walk to claudication daily.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes